CLINICAL TRIAL: NCT05846139
Title: The Effectiveness of an Incremental Approach to Nonsurgical Periodontal Therapy With the Use of Adjunctive Slow-release Locally Administered 0.02% Hypochlorite Formulation: A Single-blind Randomized Clinical Study
Brief Title: Slow-release Locally Administered 0.02% Hypochlorite Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuscan Dental Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0.02% hypochlorite formulation
Record Dates: First submitted 2023-04-16; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PerioTabs® brushing solution (Experimental): At baseline, patients were given instructions for the home use of PerioTabs® for daily gum and toothbrushing for 10 consecutive days, according to the product's directions for use. The procedure consisted of brushing the teeth and gums for 2 minutes in the evening during a 10-day period. After one week, one-stage full-mouth disinfection was performed with the use of ultrasonic devices on each quadrant. In addition, two cycles of 90 seconds ozone-therapy were carried out.
  Interventions: Combination Product: PerioTabs® brushing solution
- Chlorhexidine 0.2% mouth rinse (Active Comparator): At baseline, patients were given instructions for the home use of toothbrush with chlorhexidine 0.12 % toothpaste for 15 days toothbrushing twice daily (morning and evening). Also, a chlorhexidine 0.2% mouth rinse had to be used every evening for the course of the 15 days. After two weeks, the one-stage full-mouth disinfection was performed in the same way as in Group 1.
  Interventions: Combination Product: Chlorhexidine 0.12 %

INTERVENTIONS:
Combination Product: PerioTabs® brushing solution — PerioTabs® contains a non-antibiotic biofilm removal complex called NitrAdine®.Its anti-biofilm action is based on the combination of surfactant-induced protein denaturation and slow release of a non-toxic concentration of hypochlorite (0.02%).
  Arms: PerioTabs® brushing solution
Combination Product: Chlorhexidine 0.12 % — chlorhexidine 0.12 % toothpaste and chlorhexidine 0.2% mouth rinse
  Arms: Chlorhexidine 0.2% mouth rinse

SUMMARY:
Aim: The presence of bacterial plaque is associated with the development of periodontal inflammation. The aim of this single-blind randomized clinical study was to prospectively evaluate the efficacy of two different agents in a staged approach for nonsurgical periodontal treatment in terms of clinical and patients related outcomes in a cohort of patients with periodontitis: NitrAdine® based disinfectant formula (PerioTabs®) vs Chlorhexidine 0.12 toothpaste and mouthwash 0.20.

Material and methods: Patients with a diagnosis of periodontal disease (stage I-III) scheduled for non surgical periodontal treatment were randomly allocated to the preparatory home use of a chlorhexidine mouthwash or a NitrAdine® based brushing solution called PerioTabs® for 10-15 days. Active decontamination with ultrasonic scalers was performed after the completion of the preparation period. Clinical and patient-related outcomes were recorded at baseline, at the moment of professional intervention, and after 30 and 90 days from baseline.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 y.o,
* systemically healthy,
* with a clinical diagnosis of periodontitis

Exclusion Criteria:

* alcohol or drug abuse,
* regular drug use of bisphosphonates,
* non-steroidal or steroidal anti-inflammatory,
* daily antacid therapy,
* selective serotonin reuptake inhibitors and other therapy that might affect periodontal health,
* antibiotics during the previous 6 months,
* smoking more than ten cigarettes per day;
* pregnancy;
* lactation;
* previous periodontitis treatment within the last 6 months,
* radiotherapy to the head or neck, current chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
change in full mouth bleeding score (ΔFMBS) | Between baseline and the active debridement which occurred 15 days later

CONTACTS AND LOCATIONS:
Locations (1):
- Fortis Centro Odontoiatrico, Forte dei Marmi, Lucca, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data are available upon reasonable request from colleagues